CLINICAL TRIAL: NCT01828736
Title: Multicenter Randomized Phase 2 Trial of Gemcitabine - Platinum With or Without Trastuzumab in Advanced or Metastatic Urothelial Carcinoma With HER2 Overexpression
Brief Title: Efficacy of Combination of Trastuzumab to Gemcitabine - Platinum Advanced or Metastatic Urothelial Carcinoma
Acronym: CVH-CT02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVH-CT 02
Record Dates: First submitted 2013-04-04; First posted 2013-04-11 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Recurrent Bladder Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder
Keywords: Urothelial carcinoma; Trastuzumab; Treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Trastuzumab; Gemcitabine; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Platinum + Gemcitabine (Active Comparator): Gemcitabine = 1 000 mg/m2 Day1 and Day8 given every 21 days IV
  + If Creatinin Clearance > 60 ml/min : Cisplatin = Day 1: 70 mg/m² given every 21 days If Creatinin Clearance < 60 ml/min : Carboplatin = Day 1: AUC 5 given every 21 days
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin
- Arm B: Platinum+Gemcitabine+Trastuzumab (Experimental): Trastuzumab: Charging dose = 8mg/kg on day 1; then 6mg/kg every 21 days given IV + Gemcitabine = 1 000 mg/m2 Day1 and Day8 given every 21 days IV
  + If Creatinin Clearance > 60 ml/min : Cisplatin = Day 1: 70 mg/m² given every 21 days If Creatinin Clearance < 60 ml/min : Carboplatin = Day 1: AUC 5 given every 21 days
  Interventions: Biological: Trastuzumab; Drug: Gemcitabine; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Biological: Trastuzumab — Bottles of 150 mg; Charging dose: 8mg/kg then 6mg/kg every 21 days given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
  Arms: Arm B: Platinum+Gemcitabine+Trastuzumab
Drug: Gemcitabine — Given IV, 1000 mg/m² BSA on Day 1 and Day 8 every 21 days
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; Gemzar; gemcitabin hydrochloride
Drug: Carboplatin — Given IV: AUC 5 on Day 1 every 21 days
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: Cisplatin — Given IV, 70 mg/m² BSA on day 1 every 21 days
  Other Names: cis-Diamminedichloroplatinum(II); Platinum Diamminodichloride; Diamminodichloride, Platinum; cis-Platinum; cis Platinum; Dichlorodiammineplatinum; cis-Diamminedichloroplatinum; cis Diamminedichloroplatinum; cis-Dichlorodiammineplatinum(II); Platinol; Platidiam; Platino; NSC-119875; Biocisplatinum

SUMMARY:
A multicenter, randomized, Phase 2 trial to study the effectiveness and feasibility of association of trastuzumab with combination chemotherapy in advanced or metastatic bladder cancer patients. Combining monoclonal antibody therapy with combination chemotherapy may improve treatment efficacy on tumours overexpressed HER 2.

ELIGIBILITY:
Inclusion Criteria:

* Transitional cell carcinoma of the urothelium or bladder histologically proven stage IV AJCC [locally advanced (T4b and / or N + M0) unresectable or metastatic (M1)]
* Tumor and / or metastasis overexpressing HER2 immunohistochemistry (IHC 3 +) or IHC 2 + and FISH +. Centralized analysis.
* Measurable disease with at least one lesion with a diameter> 2 cm for conventional methods (clinical examination, CT or MRI) or> 1 cm for the helical scanner. In case of single metastasis, metastatic disease should be histologically proven
* Age ≥ 18 years and ≤80 years
* Life expectancy> 3 months,
* Index performance status <2 according to ECOG PS,
* No prior chemotherapy other than adjuvant and / or neoadjuvant chemotherapy, without Herceptin ® and complete for more than 6 months (naive to any previous chemotherapy in the metastatic setting)
* No radiotherapy within 4 weeks prior to inclusion,
* Normal cardiac function as measured by ejection fraction (LVEF> 50%),
* Blood and liver satisfactory constants:

Hematological criteria: - Neutrophils> 1.5 x 109 / L, - Chips> 100 x 109 / L - Hemoglobin> 10 g / dL, Liver function: - Alkaline phosphatase (unless bone metastases) <2 x N - Total bilirubin <1.5 x N - transaminases (AST, ALT) <1.5 x N, renal Constants: - Creatinine clearance > 30 ml / min (Cockcroft and Gault, cf. Annex XV protocol)

- Patient's written consent after full information.

Exclusion Criteria:

* Concurrent treatment with an experimental drug, participation in another clinical trial within <30 days
* Patients previously treated with Herceptin ®, or another treatment targeting growth factors EGF (eg Iressa ®, Tarceva ®)
* Existence of a severe pulmonary disease, liver or kidney is likely to be exacerbated by the treatment,
* Other medical conditions: congestive heart failure or angina pectoris even if medically controlled failure, history of myocardial infarction before entering the trial, hypertension or uncontrolled arrhythmias, significant valvular disease,
* Patient with dyspnoea at rest or requiring oxygen therapy or with respiratory failure,
* Presence of a severe infection requiring antibiotics,
* Presence of CNS metastases or meningeal
* History of another malignancy uncured or cured for less than 5 years (except basal cell carcinoma, papillary thyroid carcinoma in situ of the cervix treated)
* Pregnant or lactating or not using effective contraception Women,
* For Cisplatin only: carrying a serious neurological disease, current events devices> NCI grade 2 neuropathy, hearing loss, creatinine clearance <60 ml / min, the patient can not support a patient hydration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-02-09 (Actual); Primary Completion 2010-02-23 (Actual); Study Completion 2010-02-23 (Actual)

PRIMARY OUTCOMES:
Progression Free survival | Participants will be followed from radomization until progression or death, up to 3 years

SECONDARY OUTCOMES:
Objective response rate | Objective Response Rate will be assessed during treatment period, every 3 cycles, up to 7 months
Number of participants with adverse events as a measure of safety and tolerability | Participants will be followed all along the study period, an expected average of 3 years
  Toxicity will be classify according to NCI-CTC criteria Version 2.0. Cardiac toxicity will be assessed according to the NYHA (New York Heart Association) criteria.
Quality of life | Quality of Life will be assessed during the study period, every 3 cycles (Arm A patients) or every 3 months (Arm B patients), up to 3 years
  Quality of Life will be assessed according to the EORTC QLQ-C30 Version 3 questionnaire
Overall survival | Participants will be followed from randomization until death or lost of follow-up, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Oudard, MD, PhD., Principal Investigator — Hôpital Européen Georges Pompidou, Paris (France); Philippe Beuzeboc, MD, Principal Investigator — Curie Institute
Locations (15):
- Cliniques saint Luc - Université Catholique de Louvain, Brussels, Belgium
- France (14):
  - CHU de Besançon, Besançon
  - CHU Hôpital Saint André, Bordeaux
  - Hôpital Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Départemental de la Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - CHU Hôpital La Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Clinique Hartmann, Neuilly-sur-Seine
  - Curie Institute, Paris
  - Hôpital Saint Louis, Paris
  - Groupe Hospitalier Saint Joseph Paris, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Foch, Suresnes

REFERENCES:
- [Derived] Oudard S, Culine S, Vano Y, Goldwasser F, Theodore C, Nguyen T, Voog E, Banu E, Vieillefond A, Priou F, Deplanque G, Gravis G, Ravaud A, Vannetzel JM, Machiels JP, Muracciole X, Pichon MF, Bay JO, Elaidi R, Teghom C, Radvanyi F, Beuzeboc P. Multicentre randomised phase II trial of gemcitabine+platinum, with or without trastuzumab, in advanced or metastatic urothelial carcinoma overexpressing Her2. Eur J Cancer. 2015 Jan;51(1):45-54. doi: 10.1016/j.ejca.2014.10.009. Epub 2014 Nov 15. PMID 25459391